CLINICAL TRIAL: NCT05748938
Title: A Phase1/phase2，Single-arm, Open-label Study of RD14-01 in Patients With Advanced Solid Tumors
Brief Title: A Study of RD14-01 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD14-01-02
Record Dates: First submitted 2023-02-15; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; CAR-T Cell; ROR1
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD14-01 treated group (Experimental): Subjects who meet the enrollment conditions will receive intravenous infusion of anti--ROR1 CAR-T Cells after lymphodepleting therapy.
  Interventions: Biological: RD14-01

INTERVENTIONS:
Biological: RD14-01 — ROR1 Targeted CAR-T cells
  Other Names: CAR-T infusion

SUMMARY:
This study will evaluate the safety and tolerability of RD14-01, a ROR1-targeted CAR T-cell therapy, in patients with ROR1+ advanced solid tumors.

DETAILED DESCRIPTION:
This single-arm, open-label, dose-escalation and dose-expansion study will evaluate the safety and tolerability of RD14-01, ROR1-targeting CAR T cells, in adults with ROR1+ advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and < 70 years old, gender unlimited;
2. Patients with locally advanced or metastatic solid tumors confirmed by histopathology or cytology;
3. Subjects who failed or were intolerant to standard treatment, or lacked effective treatment;
4. ROR1+ by central laboratory immunohistochemistry (IHC);
5. Adequate organ and marrow function;
6. At least one measurable lesion as per RECIST v1.1;
7. Estimated survival ≥3 months;

7.Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1; 8.Ability to understand and provide informed consent.

Exclusion Criteria:

1. Prior treatment with any agent targeting ROR1;
2. Received anti-tumor therapy within 4 weeks prior to the start of treatment, including chemotherapy, radiotherapy, targeted therapy, etc. (excluding preconditioning);
3. Presence of active central nervous system (CNS) metastasis;
4. There is or has been a history of severe cardiovascular disease;
5. There is an uncontrolled pleural, abdominal or pericardial effusion
6. HIV-positive, active acute or chronic HBV or HCV, or active tuberculosis;
7. Pregnant or breast-feeding females;
8. There is a known or suspected failure to comply with the study protocol (for example, alcohol abuse, drug dependence, or psychological disorders) or any condition that the investigator believes may increase the subjects' risk or interfere with the results of the test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-08-08 (Estimated); Study Completion 2025-02-08 (Estimated)

PRIMARY OUTCOMES:
DLT and MTD | up to 28 days after infusion
  Dose-limiting toxicity (DLT) and maximum tolerated dose (MTD)
TEAEs | up to 12 months after infusion
  Adverse events (TEAEs) and incidence after the first infusion, treatment-related adverse events and incidence, adverse events of special concern (AESI) and incidence

SECONDARY OUTCOMES:
ORR | up to 28 days after infusion
  Overall Response Rate (ORR) by RECIST, version 1.1
DOR | up to 12 months after infusion
  Duration of response (DOR)
PFS | up to 12 months after infusion
  Progression Free Survival(PFS)
OS | up to 12 months after infusion
  Overall Survival (OS)
Maximum concentration of RD14-01 (Cmax) in peripheral blood (PB) samples | up to 12 months after infusion
  Maximum concentration of RD14-01 (Cmax) in peripheral blood (PB) samples
Persistence of RD14-01 CAR T cells in peripheral blood samples | up to 12 months after infusion
  Persistence of RD14-01 CAR T cells in peripheral blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Doctor, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China